CLINICAL TRIAL: NCT05951166
Title: Pulmonary Artery DenerVation Clinical Study Using the Gradient Denervation System in Heart Failure Patients With Pulmonary Hypertension
Acronym: PreVail-PH
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gradient Denervation Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-001
Record Dates: First submitted 2023-06-12; First posted 2023-07-18 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure Patients With Pulmonary Hypertension

STUDY DESIGN:
Intervention Model Description: A prospective, single arm, multi-center study designed to evaluate the safety, and feasibility of the Gradient Denervation System
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PADN with Gradient Denervation System (Experimental)
  Interventions: Device: Gradient Denervation System

INTERVENTIONS:
Device: Gradient Denervation System — Pulmonary artery denervation (PADN) procedure

SUMMARY:
Prospective, single-arm, multicenter First in Human study to characterize the impact of pulmonary artery denervation on the quality of life in Heart Failure Patients with Pulmonary Hypertension

ELIGIBILITY:
Inclusion Criteria:

* Heart Failure with EF ≥ 40% (by TTE within last 3 months)
* Mean Pulmonary Artery Pressure (mPAP) >20 mmHg at rest
* Pulmonary Vascular Resistance (PVR) ≥ 3WU at rest
* Pulmonary Capillary Wedge Pressure > 15 mmHg (at rest) or > 18 with passive leg raise
* Cardiac index (CI) ≥ 1.7 L/min/m2
* NYHA Class II or III
* Glomerular Filtration Rate (GFR) ≥ 25 ml/min
* N-terminal pro-B-type natriuretic peptide (NT-proBNP) ≥ 400pg/mL
* Stable, guideline directed medical treatment, including controlled volume status for a minimum of 3 months prior treatment

Exclusion Criteria:

* Inability to take dual antiplatelet or anticoagulants, hypersensitivity or allergy to aspirin or clopidogrel
* Pulmonary artery aneurysm, moderate or greater PA stenosis or other PA anatomy that would prevent safe or proper use of the study device
* Systemic infection or localized infection/rash at planned access site at time of procedure
* Myocardial infarction, unstable angina pectoris, or a cerebrovascular accident in the previous 3 months
* CRT or other Interventional cardiac procedure (except RHC) within last 3 months
* Any planned cardiac procedure or inpatient procedure within the next 30 days

Ages: 22 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-05-05 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Device related serious adverse events | 30 days post-treatment

SECONDARY OUTCOMES:
Mean change from baseline in Pulmonary Vascular Resistance (woods units) | 6- months post-treatment

CONTACTS AND LOCATIONS:
Locations (2):
- Georgia (2):
  - Israeli-Georgian Medical Research Clinic Helsicore, Tbilisi
  - Tbilisi Heart Clinic, Tbilisi

IPD SHARING:
Plan to Share IPD: No